CLINICAL TRIAL: NCT00004165
Title: Stem Cell Transplant as Standard Therapy for Symptomatic Multiple Myeloma
Brief Title: Melphalan Followed by Peripheral Stem Cell Transplantation in Treating Patients With Multiple Myeloma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: NU 97H6T; NU-97H6T; NCI-G99-1632
Record Dates: First submitted 1999-12-10; First posted 2003-01-27 (Estimated); Last update posted 2012-06-06 (Estimated); Status verified 2012-05

CONDITIONS: Multiple Myeloma and Plasma Cell Neoplasm
Keywords: refractory multiple myeloma; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; primary systemic amyloidosis
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell; Immunoglobulin Light-chain Amyloidosis | interventions — Filgrastim; Melphalan; Peripheral Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: filgrastim
Drug: melphalan
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Peripheral stem cell transplantation may allow the doctor to give higher doses of chemotherapy drugs and kill more cancer cells.

PURPOSE: Phase III trial to study the effectiveness of melphalan followed by peripheral stem cell transplantation in treating patients who have multiple myeloma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Administer standard, high dose melphalan safely in a closely monitored setting in patients with responsive multiple myeloma.
* Determine the cost and time effectiveness in the collection of sufficient peripheral blood stem cells (PBSC) for two high dose melphalan therapies and PBSC transplantations in this patient population.

OUTLINE: Patients not in remission receive 3-6 courses of remission induction therapy consisting of either an anthracycline/glucocorticoid regimen or high dose glucocorticoids.

At 21-45 days following induction therapy, patients receive filgrastim (G-CSF) subcutaneously daily for 4 days followed by daily peripheral blood stem cell (PBSC) collection beginning on day 4 and continuing until the target number of cells is reached.

At 5 days to 6 weeks following PBSC collection, patients receive high dose melphalan IV over 2 hours for 2 consecutive days. At 36-48 hours following completion of melphalan, patients receive infusion of PBSC followed by G-CSF subcutaneously daily until blood counts recover.

At 3 months to 5 years following high dose therapy and PBSC infusion, patients with evidence of disease progression receive an additional treatment with high dose melphalan followed by PBSC infusion as in the first course.

Patients are followed at 30-45 days, 6 months, and then annually thereafter.

PROJECTED ACCRUAL: A total of 60-120 patients will be accrued for this study over 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosed active multiple myeloma defined by:

  * Lytic disease
  * Anemia
  * Hypercalcemia
  * Secondary renal insufficiency
  * More than 400 mg/24 hours of urinary protein excretion
  * Symptomatic hyperviscosity
* If previously treated, refractory to no more than 1 regimen
* Primary amyloidosis without subsequent multiple myeloma allowed

  * Abnormal renal function allowed if due to primary disease

PATIENT CHARACTERISTICS:

Age:

* Not specified

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* See Disease Characteristics
* Creatinine clearance greater than 50 mL/min if no renal impairment

Cardiovascular:

* No cardiac function that would preclude study
* LVEF greater than 45%

Pulmonary:

* No pulmonary function that would preclude study
* FVC greater than 60% predicted
* DLCO greater than 50% predicted

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No greater than 18 months of prior alkylator exposure

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* See Disease Characteristics
* No more than 3 prior treatment regimens allowed

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1999-10; Primary Completion 2003-08 (Actual); Study Completion 2003-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ann Traynor, MD, Study Chair — Robert H. Lurie Cancer Center
Locations (1):
- Robert H. Lurie Comprehensive Cancer Center, Northwestern University, Chicago, Illinois, United States